CLINICAL TRIAL: NCT01394952
Title: The Effect of Dulaglutide on Major Cardiovascular Events in Patients With Type 2 Diabetes: Researching Cardiovascular Events With a Weekly INcretin in Diabetes (REWIND)
Brief Title: Researching Cardiovascular Events With a Weekly Incretin in Diabetes (REWIND)
Acronym: REWIND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13438; H9X-MC-GBDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Disease; Diabetes Mellitus, Type 2
Keywords: Cardiovascular disease; Diabetes Mellitus; Dulaglutide
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.5 mg Dulaglutide (Experimental): Administered once weekly, subcutaneously
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Administered once weekly, subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Administered subcutaneously
  Other Names: LY2189265
  Arms: 1.5 mg Dulaglutide
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess whether dulaglutide can reduce major cardiovascular events and other serious outcomes in persons with type 2 diabetes, when added to their anti-hyperglycemic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with Hemoglobin A1c equal to or less than 9.5% (equal to or less than 81 mmol/mol)
* Anti-hyperglycemic drug naive or treated with up to 2 oral hyperglycemic drugs with or without a glucagon-like peptide-1analog or basal insulin, or basal insulin alone
* On stable antihyperglycemic regimen for at least 3 months
* Age equal to or greater than 50 years with established clinical vascular disease, or age equal to or greater than 55 years and subclinical vascular disease or age equal to or greater than 60 years and at least 2 or more cardiovascular risk factors

Exclusion Criteria:

* Uncontrolled diabetes requiring immediate therapy
* History of severe hypoglycemia in past year
* Acute coronary or cerebrovascular event within past 2 months
* Planned or anticipated revascularization procedure
* History of pancreatitis, hepatic insufficiency , chronic renal failure or of C-cell thyroid disorder
* Pregnancy or planned pregnancy during the trial period
* Completed or withdrawn from any study investigating dulaglutide

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9901 (Actual)
Dates: Start 2011-07-22 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (299):
- United States (51):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pell City, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlingame, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandon, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plant City, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Charlotte, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawrenceville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalispell, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camden, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresh Meadows, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westfield, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murrells Inlet, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burke, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salem, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Argentina (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bahía Blanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cipolletti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad de Parana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coronel Suárez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corrientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Junín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merlo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rafaela Santa Fe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Nicolás
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venado Tuerto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villa María
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zárate
- Australia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milton, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clayton, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg Heights, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Brazil (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasília
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campina Grande do Sul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sao Jose Rio Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uberaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Votuporanga
- Bulgaria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Blagoevgrad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
- Canada (27):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spruce Grove, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brampton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Etobicoke, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakville, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oshawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smiths Falls, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thornhill, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fleurimont, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granby, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Laurent, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esaskatoon, Saskatchewan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
- Chile (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osomo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temuco
- Colombia (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Armenia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barranquilla
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrio Maridias
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bogotá
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cartagena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Espinal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Floridablanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manizales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medellín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pereira
- Czechia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chomutov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Havířov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinočany
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Příbram
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valašské Klobouky
- Germany (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Oeynhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dippoldiswalde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ingelheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Künzing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pirna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saarlouis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Speyer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villingen-Schwenningen
- Hungary (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kecskemét
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mosonmagyaróvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- Latvia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daugavpils
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jelgava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liepāja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limbaži
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tukums
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valmiera
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilniuslt
- Mexico (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toluca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veracruz
- New Zealand (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beckenham, Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunedin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hastings
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Papamoa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roslyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotorua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tauranga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waitakere City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westown
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puławy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sobótka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Łosice
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alba Lulia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bacau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maramures
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piteşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Satu Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sibiu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolensk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Volgograd
- South Africa (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benoni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Die Wilgers Ext 14
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grassy Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lynnwood Ridge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyttleton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rondebosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Soweto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tongaat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guri-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Centelles
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Segovia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vic
- Sweden (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aneby
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Härnösand
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Köping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ljungby
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Östersund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skellefteå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vaxjo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vällingby
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung Hsien
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
- United Kingdom (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlesbrough, Cleveland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hull, East Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldham, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belfast, Northern Ireland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ayr, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inverness, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swansea, Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antrim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belfast
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Londonderry

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Gerstein HC, Lee SF, Pare G, Bethel MA, Colhoun HM, Hoover A, Lakshmanan M, Lin Y, Pirro V, Qian HR, Ruotolo G, Ryden L, Wilson JM, Duffin KL. Biomarker Changes Associated With Both Dulaglutide and Cardiovascular Events in the REWIND Randomized Controlled Trial: A Nested Case-Control Post Hoc Analysis. Diabetes Care. 2023 May 1;46(5):1046-1051. doi: 10.2337/dc22-2397. PMID 36897834
- [Derived] Ferrannini G, Maldonado JM, Raha S, Rao-Melacini P, Khatun R, Atisso C, Shurzinske L, Gerstein HC, Ryden L, Bethel MA. Gender differences in cardiovascular risk, treatment, and outcomes: a post hoc analysis from the REWIND trial. Scand Cardiovasc J. 2023 Dec;57(1):2166101. doi: 10.1080/14017431.2023.2166101. PMID 36723445
- [Derived] Gerstein HC, Ramasundarahettige C, Avezum A, Basile J, Conget I, Cushman WC, Dagenais GR, Franek E, Lakshmanan M, Lanas F, Leiter LA, Pogosova N, Probstfield J, Raubenheimer PJ, Riddle M, Shaw J, Sheu WH, Temelkova-Kurktschiev T, Turfanda I, Xavier D. A novel kidney disease index reflecting both the albumin-to-creatinine ratio and estimated glomerular filtration rate, predicted cardiovascular and kidney outcomes in type 2 diabetes. Cardiovasc Diabetol. 2022 Aug 22;21(1):158. doi: 10.1186/s12933-022-01594-6. PMID 35996147
- [Derived] Franek E, Gerstein HC, Riddle MC, Nicolay C, Hickey A, Botros FT, Loo LS. Efficacy and safety outcomes of dulaglutide by baseline HbA1c: A post hoc analysis of the REWIND trial. Diabetes Obes Metab. 2022 Sep;24(9):1753-1761. doi: 10.1111/dom.14760. Epub 2022 May 30. PMID 35546279
- [Derived] Cukierman-Yaffe T, Gerstein HC, Basile J, Bethel MA, Cardona-Munoz EG, Conget I, Dagenais G, Franek E, Hall S, Hancu N, Jansky P, Lakshmanan M, Lanas F, Leiter LA, Lopez-Jaramillo P, Pirags V, Pogosova N, Probstfield J, Rao-Melacini P, Ramasundarahettige C, Raubenheimer PJ, Riddle MC, Ryden L, Shaw JE, Sheu WH, Temelkova-Kurktschiev T. Novel Indices of Cognitive Impairment and Incident Cardiovascular Outcomes in the REWIND Trial. J Clin Endocrinol Metab. 2022 Jul 14;107(8):e3448-e3454. doi: 10.1210/clinem/dgac200. PMID 35446415
- [Derived] Kwan AYM, Gerstein HC, Basile J, Xavier D, Maldonado JM, Raha S, Konig M. HbA1c Reduction in Dulaglutide-Treated Patients Irrespective of Duration of Diabetes, Microvascular Disease, and BMI: A Post Hoc Analysis From the REWIND Trial. Diabetes Care. 2022 Mar 1;45(3):547-554. doi: 10.2337/dc21-1160. PMID 35043140
- [Derived] Konig M, Riddle MC, Colhoun HM, Branch KR, Atisso CM, Lakshmanan MC, Mody R, Raha S, Gerstein HC. Exploring potential mediators of the cardiovascular benefit of dulaglutide in type 2 diabetes patients in REWIND. Cardiovasc Diabetol. 2021 Sep 25;20(1):194. doi: 10.1186/s12933-021-01386-4. PMID 34563178
- [Derived] Bajaj HS, Gerstein HC, Rao-Melacini P, Basile J, Colhoun H, Conget I, Cushman WC, Dagenais GR, Franek E, Hanefeld M, Keltai M, Lakshmanan M, Lanas F, Leiter LA, Lopez-Jaramillo P, Pirags V, Pogosova N, Probstfield J, Raubenheimer P, Ryden L, Shaw JE, Sheu WH, Xavier D. Erectile function in men with type 2 diabetes treated with dulaglutide: an exploratory analysis of the REWIND placebo-controlled randomised trial. Lancet Diabetes Endocrinol. 2021 Aug;9(8):484-490. doi: 10.1016/S2213-8587(21)00115-7. Epub 2021 Jun 18. PMID 34153269
- [Derived] Riddle MC, Gerstein HC, Xavier D, Cushman WC, Leiter LA, Raubenheimer PJ, Atisso CM, Raha S, Varnado OJ, Konig M, Lakshmanan M, Franek E. Efficacy and Safety of Dulaglutide in Older Patients: A post hoc Analysis of the REWIND trial. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1345-1351. doi: 10.1210/clinem/dgab065. PMID 33537745
- [Derived] Dagenais GR, Ryden L, Leiter LA, Lakshmanan M, Dyal L, Probstfield JL, Atisso CM, Shaw JE, Conget I, Cushman WC, Lopez-Jaramillo P, Lanas F, Munoz EGC, Pirags V, Pogosova N, Basile J, Sheu WHH, Temelkova-Kurktschiev T, Raubenheimer PJ, Keltai M, Hall S, Pais P, Colhoun HM, Riddle MC, Gerstein HC. Total cardiovascular or fatal events in people with type 2 diabetes and cardiovascular risk factors treated with dulaglutide in the REWIND trail: a post hoc analysis. Cardiovasc Diabetol. 2020 Nov 25;19(1):199. doi: 10.1186/s12933-020-01179-1. PMID 33239067
- [Derived] Cukierman-Yaffe T, Gerstein HC, Colhoun HM, Diaz R, Garcia-Perez LE, Lakshmanan M, Bethel A, Xavier D, Probstfield J, Riddle MC, Ryden L, Atisso CM, Hall S, Rao-Melacini P, Basile J, Cushman WC, Franek E, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T. Effect of dulaglutide on cognitive impairment in type 2 diabetes: an exploratory analysis of the REWIND trial. Lancet Neurol. 2020 Jul;19(7):582-590. doi: 10.1016/S1474-4422(20)30173-3. PMID 32562683
- [Derived] Gerstein HC, Hart R, Colhoun HM, Diaz R, Lakshmanan M, Botros FT, Probstfield J, Riddle MC, Ryden L, Atisso CM, Dyal L, Hall S, Avezum A, Basile J, Conget I, Cushman WC, Hancu N, Hanefeld M, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Munoz EGC, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T. The effect of dulaglutide on stroke: an exploratory analysis of the REWIND trial. Lancet Diabetes Endocrinol. 2020 Feb;8(2):106-114. doi: 10.1016/S2213-8587(19)30423-1. Epub 2020 Jan 7. PMID 31924562
- [Derived] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Derived] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Botros FT, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and renal outcomes in type 2 diabetes: an exploratory analysis of the REWIND randomised, placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):131-138. doi: 10.1016/S0140-6736(19)31150-X. Epub 2019 Jun 9. PMID 31189509
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361
- [Derived] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riddle MC, Ryden L, Xavier D, Atisso CM, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona-Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw J, Sheu WH, Temelkova-Kurktschiev T; REWIND Trial Investigators. Design and baseline characteristics of participants in the Researching cardiovascular Events with a Weekly INcretin in Diabetes (REWIND) trial on the cardiovascular effects of dulaglutide. Diabetes Obes Metab. 2018 Jan;20(1):42-49. doi: 10.1111/dom.13028. Epub 2017 Jul 14. PMID 28573765

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to either placebo or Dulaglutide. Completers included participants for whom vital status was ascertained during the study close-out period and endpoint completers.
Groups:
- Placebo: Placebo was administered once weekly, subcutaneously
- Dulaglutide: 1.5 mg Dulaglutide was administered once weekly, subcutaneously
Period: Overall Study
Arm/Group | Placebo | Dulaglutide
Started | 4952 | 4949
Received at Least One Dose of Study Drug | 4949 | 4943
Completed | 4935 | 4932
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 0 | 5
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor Decision | 5 | 7

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dulaglutide | Total
Number analyzed (Participants) | 4952 | 4949 | 9901
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2315 | 2330 | 4645
  >=65 years | 2637 | 2619 | 5256
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.5) | 66.2 (6.5) | 66.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2283 | 2306 | 4589
  Male | 2669 | 2643 | 5312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 60 | 124
  Not Hispanic or Latino | 402 | 400 | 802
  Unknown or Not Reported | 4486 | 4489 | 8975
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 543 | 549 | 1092
  Asian | 218 | 216 | 434
  Native Hawaiian or Other Pacific Islander | 22 | 12 | 34
  Black or African American | 346 | 331 | 677
  White | 3744 | 3754 | 7498
  More than one race | 79 | 87 | 166
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Puerto Rico is combined with the United States for this study.
  Participants
    United States | 475 | 468 | 943
    Czechia | 107 | 106 | 213
    Russia | 50 | 51 | 101
    South Korea | 62 | 60 | 122
    Sweden | 117 | 119 | 236
    Latvia | 39 | 39 | 78
    Brazil | 137 | 138 | 275
    Poland | 305 | 303 | 608
    Chile | 64 | 64 | 128
    Bulgaria | 50 | 51 | 101
    Lithuania | 52 | 53 | 105
    Colombia | 392 | 393 | 785
    Argentina | 698 | 697 | 1395
    Romania | 544 | 541 | 1085
    Hungary | 113 | 110 | 223
    United Kingdom | 65 | 71 | 136
    Spain | 62 | 65 | 127
    New Zealand | 119 | 115 | 234
    Canada | 564 | 564 | 1128
    Taiwan | 13 | 13 | 26
    South Africa | 369 | 372 | 741
    Mexico | 219 | 219 | 438
    Australia | 44 | 44 | 88
    Germany | 292 | 293 | 585

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Event For Time, From Randomization to First Occurrence of Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke (a Composite Cardiovascular Outcome)
Description: The time from randomization to first occurrence of cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke (a composite endpoint) was evaluated using time-to-event analysis. The primary analysis model was a Cox proportional hazards regression model for the time to the first occurrence of a primary endpoint event, with treatment as a fixed effect using the intent-to-treat population. The number of participants who experienced a primary cardiovascular (CV) endpoint event is presented.
Time Frame: From randomization to first occurrence or death from any cause or study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants | 663 | 594
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Primary CV endpoint; Test type: Superiority — Superiority was declared if the upper limit of the 2-sided 95.33% confidence interval (CI) of the hazard ratio was below 1.0 (after adjustment for the interim analysis). Once superiority was achieved for the primary endpoint, multiplicity adjustments using the graphical approach were performed for secondary efficacy endpoints in order to control the overall Type I error rate at a 2-sided alpha level of 0.0467; p = 0.026, Regression, Cox; Hazard Ratio (HR) = 0.88, 95.33% CI 2-sided [0.79 to 0.99]

2. Secondary Outcome: Number of Participants Who Experienced an Event for Time to First Occurrence After Randomization of Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke, Individually
Description: The time from randomization to first occurrence of cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke (individually) was evaluated using time-to-event analysis via the Cox proportional hazards regression model where response equals treatment. Death from CV causes is defined as a death resulting from an acute myocardial infarction (MI), sudden cardiac death, death due to heart failure, death due to stroke, or death due to other CV causes. The number of participants who experienced an event is presented.
Time Frame: From randomization to first occurrence or study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants
  Death from CV causes | 346 | 317
  Nonfatal MI | 212 | 205
  Nonfatal stroke | 175 | 135
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Death from CV causes; Test type: Superiority — Multiplicity adjustments using the graphical approach were performed for secondary efficacy endpoints in order to control the overall Type I error rate at a 2-sided alpha level of 0.0467; p = 0.211, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.78 to 1.06]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide; Nonfatal MI; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.652, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.79 to 1.16]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide; Nonfatal stroke; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.017, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.61 to 0.95]

3. Secondary Outcome: Number of Participants Who Experienced an Event for Time to All-cause Mortality
Description: The time to all-cause mortality was evaluated using time-to-event analysis via the Cox proportional hazards regression model where response equals treatment. The number of participants who experienced an event is presented.
Time Frame: From randomization to study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants | 592 | 536
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Time to all cause mortality; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.067, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.80 to 1.01]

4. Secondary Outcome: Number of Participants Who Experienced an Event for Time to First Occurrence After Randomization of the Composite Microvascular Endpoint
Description: The time from randomization to first occurrence of the composite microvascular endpoint was evaluated using time-to-event analysis via the Cox proportional hazards regression model where response equals treatment. The composite microvascular endpoint is defined as diabetic retinopathy requiring laser therapy, vitrectomy, or anti-vascular endothelial growth factor therapy (VEGF), clinical proteinuria, a greater than equal ≥ 30% decline in estimated glomerular filtration rate, or need for chronic renal replacement therapy. The number of participants who experienced the composite microvascular endpoint event is presented.
Time Frame: From randomization to first occurrence or study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants | 1241 | 1099
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; microvascular endpoint; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.79 to 0.93]

5. Secondary Outcome: Number of Participants Who Experienced An Event for Time to First Occurrence After Randomization of Heart Failure Requiring Hospitalization or an Urgent Heart Failure Clinic Visit
Description: The time to first occurrence after randomization of heart failure requiring hospitalization or an urgent heart failure clinic visit was evaluated using time-to-event analysis via the Cox proportional hazards regression model where response equals treatment. The number of participants who experienced an event is presented.
Time Frame: From randomization to first occurrence or study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants | 226 | 213
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Heart failure requiring hospitalization or an urgent heart failure clinic visit; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.456, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.12]

6. Secondary Outcome: Number of Participants Who Experienced an Event for Time to First Occurrence After Randomization of First Hospitalization for Unstable Angina
Description: Time to first occurrence after randomization of first hospitalization for unstable angina was evaluated using time-to-event analysis via the Cox proportional hazards regression model where response equals treatment. The number of participants who experienced an event is presented.
Time Frame: From randomization to first occurrence or study completion (Median Follow-Up of 5.4 Years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dulaglutide
Number analyzed (Participants) | 4952 | 4949
Participants | 77 | 88
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide; Hospitalization for unstable angina; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.413, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.84 to 1.54]

ADVERSE EVENTS:
Time Frame: From Randomization to Study Completion (Up to 7 Years)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Placebo | Dulaglutide
All-Cause Mortality (participants affected / at risk) | 592/4949 | 536/4943
Serious Adverse Events (participants affected / at risk) | 2044/4949 | 1991/4943
Other Adverse Events (participants affected / at risk) | 3363/4949 | 3574/4943
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=4949) | Dulaglutide (N=4943)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 23 (24) | 29 (30)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (10) | 14 (14)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 41 (43) | 43 (44)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 53 (59) | 39 (40)
Angina pectoris (Cardiac disorders) | 58 (67) | 56 (61)
Angina unstable (Cardiac disorders) | 54 (58) | 44 (47)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 5 (5)
Aortic valve stenosis (Cardiac disorders) | 6 (7) | 9 (9)
Arrhythmia (Cardiac disorders) | 3 (3) | 6 (6)
Arteriosclerosis coronary artery (Cardiac disorders) | 9 (9) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 62 (79) | 90 (107)
Atrial flutter (Cardiac disorders) | 18 (19) | 15 (19)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 6 (6) | 7 (7)
Atrioventricular block complete (Cardiac disorders) | 11 (12) | 8 (8)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 9 (9) | 8 (8)
Bifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 3 (3) | 3 (3)
Bradycardia (Cardiac disorders) | 10 (10) | 16 (17)
Bundle branch block left (Cardiac disorders) | 3 (3) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 14 (15) | 11 (14)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 104 (124) | 78 (87)
Cardiac failure acute (Cardiac disorders) | 9 (10) | 8 (11)
Cardiac failure chronic (Cardiac disorders) | 21 (24) | 14 (15)
Cardiac failure congestive (Cardiac disorders) | 47 (52) | 38 (42)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 7 (7) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 5 (5)
Cardiomyopathy (Cardiac disorders) | 5 (5) | 2 (2)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 3 (3) | 7 (7)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 57 (64) | 57 (63)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 5 (5)
Defect conduction intraventricular (Cardiac disorders) | 2 (2) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Gastrocardiac syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 10 (11)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 8 (8) | 13 (13)
Metabolic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (3) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 7 (7) | 9 (9)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 35 (37) | 30 (30)
Myocardial ischaemia (Cardiac disorders) | 23 (23) | 19 (20)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2)
Pericarditis (Cardiac disorders) | 6 (6) | 2 (3)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 1 (2)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 6 (6) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 9 (9) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 9 (9) | 7 (7)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (4)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 5 (10) | 7 (11)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chronic granulomatous disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital cerebrovascular anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Exomphalos (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Hereditary motor and sensory neuropathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0/2667 (0) | 2/2640 (2)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1/2667 (1) | 3/2640 (3)
Vascular malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Acromegaly (Endocrine disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 8 (8) | 12 (12)
Hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hypoparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Parathyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Primary hyperaldosteronism (Endocrine disorders) | 0 (0) | 1 (2)
Thyroid mass (Endocrine disorders) | 2 (2) | 2 (2)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Blepharochalasis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 29 (34) | 19 (27)
Cataract diabetic (Eye disorders) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 3 (4) | 0 (0)
Cataract subcapsular (Eye disorders) | 2 (2) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 2 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (8) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (3) | 0 (0)
Glaucoma (Eye disorders) | 6 (6) | 3 (3)
Hypermetropia (Eye disorders) | 1 (2) | 0 (0)
Iridodialysis (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 2 (2)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 1 (1)
Maculopathy (Eye disorders) | 1 (2) | 0 (0)
Neurotrophic keratopathy (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 2 (3) | 0 (0)
Ophthalmic vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 1 (1) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 3 (4)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 3 (4)
Abdominal adhesions (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 7 (7) | 7 (7)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 10 (12)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 2 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 7 (9) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 4 (4)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 10 (10)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enteritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (3) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gallstone ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 7 (7) | 6 (6)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (3) | 8 (8)
Gastritis (Gastrointestinal disorders) | 17 (17) | 13 (13)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (14) | 12 (13)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal mucocoele (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 9 (9)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 5 (5)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Heyde's syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 7 (7)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 11 (11) | 17 (17)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 14 (15) | 9 (9)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (3) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 4 (6)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 6 (6)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 3 (3) | 2 (2)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Necrotising oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Palatal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 9 (9)
Pancreatitis acute (Gastrointestinal disorders) | 8 (10) | 15 (15)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal venous gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 5 (5)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (12) | 5 (5)
Spigelian hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 7 (7) | 3 (3)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (10) | 7 (7)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (3)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (8)
Adverse drug reaction (General disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 5 (5) | 5 (6)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 14 (15) | 7 (7)
Death (General disorders) | 9 (9) | 9 (9)
Device intolerance (General disorders) | 1 (1) | 0 (0)
Drug effect increased (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 4 (4)
Generalised oedema (General disorders) | 4 (4) | 2 (2)
Hernia perforation (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 5 (5) | 4 (4)
Inflammation (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Metaplasia (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 5 (5)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 37 (44) | 26 (28)
Oedema peripheral (General disorders) | 7 (7) | 4 (4)
Pain (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 7 (7)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 5 (5) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 2 (2)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 7 (7) | 8 (8)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary dyspepsia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 6 (6)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholangitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 15 (15) | 25 (28)
Cholecystitis acute (Hepatobiliary disorders) | 17 (17) | 26 (27)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 7 (7)
Cholelithiasis (Hepatobiliary disorders) | 49 (51) | 42 (43)
Cholestasis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 1 (1)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 2 (2)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 4 (4) | 5 (5)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Immunodeficiency (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 3 (4) | 3 (4)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 4 (4) | 4 (4)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Aortitis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 6 (6)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 4 (4) | 1 (1)
Arthritis infective (Infections and infestations) | 4 (4) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 6 (6) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 12 (12) | 13 (13)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Candida sepsis (Infections and infestations) | 1 (1) | 1 (1)
Candiduria (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 42 (48) | 38 (39)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Cervicitis (Infections and infestations) | 0/2282 (0) | 1/2303 (1)
Cholecystitis infective (Infections and infestations) | 2 (2) | 2 (2)
Chronic hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 5 (6)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 2 (2)
Corneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 6 (6) | 3 (3)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 3 (3) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) | 3 (6)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 5 (5) | 1 (1)
Diabetic gangrene (Infections and infestations) | 3 (3) | 1 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 10 (12) | 15 (17)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Echinococciasis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 4 (5)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0/2667 (0) | 4/2640 (4)
Erysipelas (Infections and infestations) | 15 (18) | 11 (12)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder abscess (Infections and infestations) | 2 (2) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 11 (11) | 8 (18)
Gastroenteritis (Infections and infestations) | 10 (10) | 21 (22)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 3 (3) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis c (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis e (Infections and infestations) | 1 (2) | 0 (0)
Hepatitis infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (5) | 0 (0)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Hydrocele male infected (Infections and infestations) | 0/2667 (0) | 1/2640 (1)
Implant site infection (Infections and infestations) | 0 (0) | 2 (2)
Infected skin ulcer (Infections and infestations) | 3 (3) | 4 (4)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 6 (8) | 3 (3)
Influenza (Infections and infestations) | 8 (8) | 5 (5)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (2) | 1 (1)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 2 (2) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 4 (4)
Localised infection (Infections and infestations) | 8 (8) | 8 (8)
Lower respiratory tract infection (Infections and infestations) | 11 (12) | 12 (13)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Myiasis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 2 (2) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 2/2667 (2) | 3/2640 (3)
Osteomyelitis (Infections and infestations) | 11 (13) | 10 (11)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 2 (2)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 2 (2)
Pelvic abscess (Infections and infestations) | 1 (1) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 2 (2) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 3 (3)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 151 (174) | 135 (152)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 2 (2) | 3 (3)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 2 (2)
Postoperative abscess (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 7 (7)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 4 (4)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 15 (15) | 8 (8)
Pyelonephritis acute (Infections and infestations) | 8 (8) | 7 (7)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 1 (1)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1/2667 (1) | 0/2640 (0)
Sepsis (Infections and infestations) | 35 (37) | 30 (33)
Septic shock (Infections and infestations) | 22 (24) | 15 (16)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin graft infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 3 (3)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (3)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 2 (3) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 61 (65) | 64 (78)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 19 (20) | 24 (26)
Vestibular neuronitis (Infections and infestations) | 3 (3) | 4 (4)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 5 (5) | 1 (1)
Wound sepsis (Infections and infestations) | 3 (3) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 20 (20) | 21 (21)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 124 (137) | 110 (123)
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 21 (22) | 18 (18)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 17 (17) | 12 (12)
Humerus fracture (Injury, poisoning and procedural complications) | 20 (20) | 12 (12)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (7) | 6 (6)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (6) | 5 (5)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 4 (4) | 12 (12)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Multiple injuries (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 7 (7)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Rib fracture (Injury, poisoning and procedural complications) | 14 (14) | 10 (10)
Road traffic accident (Injury, poisoning and procedural complications) | 9 (10) | 13 (13)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Sciatic nerve injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1/2667 (1) | 0/2640 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Subdural haematoma (Injury, poisoning and procedural complications) | 7 (7) | 7 (8)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Tibia fracture (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 3 (3)
Blood glucose increased (Investigations) | 4 (4) | 5 (6)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 2 (2)
Troponin t increased (Investigations) | 0 (0) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 14 (15) | 23 (24)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 67 (75) | 46 (52)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (12) | 8 (9)
Hyperosmolar state (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 72 (80) | 62 (69)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (12) | 8 (8)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Articular calcification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 6 (6)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Chondropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diabetic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 21 (22) | 15 (16)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 11 (14) | 10 (10)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 110 (128) | 136 (155)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 10 (11) | 8 (8)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (13)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 (23) | 16 (19)
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11) | 7 (7)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 17 (17)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 1/2303 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 7 (7)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 1/2303 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 11 (11)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 1/2303 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2282 (2) | 4/2303 (4)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2282 (2) | 0/2303 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 4 (4)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 5 (5)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Diffuse large b-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9/2282 (9) | 6/2303 (7)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 3/2303 (3)
Extranodal marginal zone b-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 7 (7)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liposarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (7)
Lung adenocarcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 9 (9)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Malignant joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Malignant melanoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2667 (0) | 3/2640 (3)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2282 (2) | 0/2303 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2282 (2) | 0/2303 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 0/2303 (0)
Ovarian cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 0/2303 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 2/2303 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (8)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2667 (1) | 0/2640 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (6)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33/2667 (34) | 33/2640 (33)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/2667 (4) | 2/2640 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2667 (1) | 1/2640 (1)
Prostate cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2667 (1) | 0/2640 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/2667 (3) | 6/2640 (6)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 3 (3)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 1/2303 (1)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 1/2303 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2282 (0) | 2/2303 (2)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2282 (2) | 4/2303 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 3/2303 (3)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2282 (1) | 1/2303 (1)
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acoustic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Amputation stump pain (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 3 (3)
Ataxia (Nervous system disorders) | 2 (2) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 4 (4) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 9 (10) | 5 (5)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 5 (5) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 4 (4) | 5 (5)
Cerebral ischaemia (Nervous system disorders) | 4 (4) | 5 (5)
Cerebrovascular accident (Nervous system disorders) | 31 (34) | 24 (25)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular insufficiency (Nervous system disorders) | 3 (3) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 3 (3) | 2 (2)
Coma (Nervous system disorders) | 0 (0) | 2 (2)
Dementia (Nervous system disorders) | 2 (2) | 4 (4)
Dementia alzheimer's type (Nervous system disorders) | 2 (2) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 8 (8) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 9 (9)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (4)
Epilepsy (Nervous system disorders) | 8 (8) | 1 (1)
Facial paralysis (Nervous system disorders) | 3 (3) | 5 (5)
Frontal lobe epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (2)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 3 (3)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hemiparesis (Nervous system disorders) | 5 (5) | 1 (1)
Hemiplegia (Nervous system disorders) | 2 (2) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 4 (6) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Iiird nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 2 (3)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Ischaemic stroke (Nervous system disorders) | 18 (22) | 14 (15)
Lacunar infarction (Nervous system disorders) | 1 (1) | 3 (3)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Language disorder (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 3 (3)
Lumbar radiculopathy (Nervous system disorders) | 4 (4) | 2 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 5 (5)
Migraine (Nervous system disorders) | 0 (0) | 2 (3)
Mixed dementia (Nervous system disorders) | 1 (1) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1) | 1 (1)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 3 (3) | 0 (0)
Myelopathy (Nervous system disorders) | 2 (2) | 2 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 5 (5)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 2 (2)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 1 (1)
Partial seizures (Nervous system disorders) | 3 (3) | 2 (3)
Peripheral nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 2 (3) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 4 (4)
Pseudobulbar palsy (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Quadriplegia (Nervous system disorders) | 0 (0) | 3 (3)
Radiculopathy (Nervous system disorders) | 3 (3) | 1 (1)
Sciatica (Nervous system disorders) | 7 (8) | 6 (6)
Seizure (Nervous system disorders) | 5 (5) | 7 (7)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 33 (34) | 36 (38)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 23 (24) | 22 (25)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 4 (4) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Vascular parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 2 (2)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Device damage (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 4 (4) | 0 (0)
Device failure (Product Issues) | 4 (4) | 1 (1)
Device loosening (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 7 (7) | 9 (9)
Delirium (Psychiatric disorders) | 8 (10) | 10 (10)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 7 (8) | 6 (6)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 3 (3)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Somatic delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 67 (74) | 61 (72)
Atonic urinary bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder dysfunction (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder fibrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 1 (2)
Bladder neck sclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 5 (5)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 19 (20) | 13 (13)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 5 (5) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 6 (6) | 3 (3)
Haematuria (Renal and urinary disorders) | 7 (8) | 2 (2)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Kidney perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 17 (18) | 18 (19)
Nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 6 (7) | 7 (8)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 17 (17) | 16 (16)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal impairment (Renal and urinary disorders) | 6 (6) | 7 (8)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 2 (2) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 9 (10) | 9 (9)
Urethral caruncle (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 4 (4) | 4 (5)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 9 (9) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 18/2667 (20) | 21/2640 (21)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 1/2282 (1) | 2/2303 (2)
Cystocele (Reproductive system and breast disorders) | 4/2282 (5) | 3/2303 (4)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/2282 (0) | 1/2303 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0/2282 (0) | 1/2303 (1)
Endometriosis (Reproductive system and breast disorders) | 0/2282 (0) | 1/2303 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1/2667 (1) | 0/2640 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0/2282 (0) | 2/2303 (3)
Fibrocystic breast disease (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Gynaecomastia (Reproductive system and breast disorders) | 0/2667 (0) | 2/2640 (3)
Metrorrhagia (Reproductive system and breast disorders) | 0/2282 (0) | 2/2303 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1/2282 (1) | 6/2303 (6)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 2/2667 (2) | 0/2640 (0)
Prostatitis (Reproductive system and breast disorders) | 2/2667 (2) | 4/2640 (4)
Prostatomegaly (Reproductive system and breast disorders) | 1/2667 (1) | 0/2640 (0)
Rectocele (Reproductive system and breast disorders) | 1/2282 (1) | 1/2303 (1)
Uterine disorder (Reproductive system and breast disorders) | 0/2282 (0) | 1/2303 (1)
Uterine polyp (Reproductive system and breast disorders) | 2/2282 (2) | 3/2303 (3)
Uterine prolapse (Reproductive system and breast disorders) | 0/2282 (0) | 3/2303 (3)
Uterovaginal prolapse (Reproductive system and breast disorders) | 2/2282 (2) | 2/2303 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/2282 (1) | 1/2303 (1)
Vaginal polyp (Reproductive system and breast disorders) | 1/2282 (1) | 0/2303 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0/2282 (0) | 2/2303 (2)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 6 (7)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 8 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 35 (45) | 25 (32)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 11 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (14)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 13 (13)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 22 (23)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 6 (6)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 16 (16)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 19 (24) | 14 (17)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 15 (16) | 9 (13)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diet noncompliance (Social circumstances) | 1 (1) | 0 (0)
Organ donor (Social circumstances) | 0 (0) | 1 (1)
Angiodysplasia (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2) | 10 (10)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 16 (17) | 21 (21)
Arterial occlusive disease (Vascular disorders) | 3 (4) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 6 (6) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 10 (10) | 16 (16)
Dry gangrene (Vascular disorders) | 2 (2) | 3 (3)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 3 (4) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 4 (4)
Haemodynamic instability (Vascular disorders) | 1 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 27 (29) | 22 (24)
Hypertensive crisis (Vascular disorders) | 21 (21) | 14 (14)
Hypertensive emergency (Vascular disorders) | 3 (3) | 4 (4)
Hypotension (Vascular disorders) | 7 (7) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 4 (4) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (2) | 0 (0)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 6 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 25 (26) | 17 (18)
Peripheral artery occlusion (Vascular disorders) | 4 (4) | 8 (9)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 8 (9) | 9 (13)
Peripheral vascular disorder (Vascular disorders) | 7 (8) | 8 (8)
Peripheral venous disease (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 3 (3)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Varicose vein (Vascular disorders) | 4 (4) | 3 (3)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=4949) | Dulaglutide (N=4943)
Cataract (Eye disorders) | 368 (417) | 363 (427)
Constipation (Gastrointestinal disorders) | 208 (223) | 361 (409)
Diarrhoea (Gastrointestinal disorders) | 436 (546) | 665 (843)
Dyspepsia (Gastrointestinal disorders) | 147 (150) | 291 (331)
Nausea (Gastrointestinal disorders) | 269 (310) | 735 (968)
Vomiting (Gastrointestinal disorders) | 154 (165) | 325 (498)
Bronchitis (Infections and infestations) | 421 (554) | 408 (528)
Influenza (Infections and infestations) | 404 (488) | 369 (435)
Nasopharyngitis (Infections and infestations) | 535 (771) | 564 (800)
Upper respiratory tract infection (Infections and infestations) | 407 (589) | 368 (533)
Urinary tract infection (Infections and infestations) | 517 (749) | 545 (795)
Decreased appetite (Metabolism and nutrition disorders) | 104 (109) | 325 (379)
Hyperglycaemia (Metabolism and nutrition disorders) | 315 (445) | 158 (190)
Hypoglycaemia (Metabolism and nutrition disorders) | 354 (1160) | 413 (1477)
Arthralgia (Musculoskeletal and connective tissue disorders) | 389 (469) | 371 (446)
Back pain (Musculoskeletal and connective tissue disorders) | 416 (484) | 447 (494)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 318 (373) | 329 (372)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 245 (280) | 260 (296)
Dizziness (Nervous system disorders) | 296 (339) | 318 (373)
Headache (Nervous system disorders) | 288 (382) | 324 (414)
Microalbuminuria (Renal and urinary disorders) | 259 (263) | 232 (241)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 135/2667 (137) | 140/2640 (144)
Cough (Respiratory, thoracic and mediastinal disorders) | 256 (292) | 239 (265)
Hypertension (Vascular disorders) | 432 (491) | 345 (405)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT01394952/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT01394952/SAP_001.pdf